CLINICAL TRIAL: NCT03548974
Title: Internet-based Physical Activity Promotion Using the MOTOmed Movement Trainer to Reduce Spasticity and Improve Physical Function in Moderately to Severely Affected Persons With Multiple Sclerosis
Brief Title: Internet-based MOTOmed Exercise to Reduce Spasticity and Improve Physical Function in Persons With Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Erlangen-Nürnberg (Other)
Collaborators: Fa. Reck MOTOmed (Unknown)
Responsible Party: Principal Investigator, Prof. Dr. Klaus Pfeifer, Prof. Dr., University of Erlangen-Nürnberg
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ATRT-2015
Record Dates: First submitted 2017-11-02; First posted 2018-06-07 (Actual); Last update posted 2018-06-07 (Actual); Status verified 2018-05

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Spasticity; MOTOmed training; internet
MeSH Terms: conditions — Multiple Sclerosis; Muscle Spasticity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Interventiongroup1 (Active Comparator): passive, motor-driven movement therapy followed by intermittent active and passive training
  Interventions: Behavioral: Treatment group 1
- Interventiongroup2 (Active Comparator): intermittent active and passive training followed by no intervention
  Interventions: Behavioral: Treatment group 2

INTERVENTIONS:
Behavioral: Treatment group 1 — The ms-intakt/MOTOmed-intervention is a home-based program using the MOTOmed movement trainer: 12 week passive, motor-driven movement therapy followed by 12 weeks of intermittent active and passive training after the 3month assessment. Training intensity was regulated by the participant's subjective, perceived exertion, which was rated between 6 and 20 on the BORG Scale. Therapists aimed at eliciting a BORG Feedback of between 10 (fairly light) and 15 (hard). The exercise training was home-based and supervised via the internet.
  Arms: Interventiongroup1
Behavioral: Treatment group 2 — The subjects assigned to interventiongroup2 started with 12 weeks intermittent active and passive training followed by 12 weeks of no intervention (Wash out phase)
  Arms: Interventiongroup2

SUMMARY:
In an RCT, the effect of the MOTOmed movement trainer (Reck, Germany) on spasticity and physical function in pwMS with EDSS score between 4,5 and 7 is investigated. All subjects exercise at home and are supervised and supported by an exercise therapist via an online platform.

We compare the effect of a 12 week passive, motor-driven movement therapy (VG1) to an intermittent active and passive training (VG2). After 12 weeks, VG1 continues with an active training including strengthening exercises for another 12 weeks. VG2 does not receive any intervention in the second study phase.

ELIGIBILITY:
Inclusion Criteria:

diagnosed Multiple Sclerosis (McDonald criteria) EDSS score between 5,5 and 7 diagnosed spasticity access to the internet

Exclusion Criteria:

lack of medical certificate for physical activity cognitive impairment clinically relevant internal disease, especially cardiovascular or pulmonary disease, metabolic and orthopedic diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2015-01; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Change in spasticity: MSSS-88 | Assessments took place at baseline, at 3 and 6 months
  This questionnaire contains 88 items, which represent the impairment by the spasticity in various subscales. The total score ranges from 88 to a maximum of 352 points (maximum impairment).
Change in sSpasticity: Modified Tardieu scale | Assessments took place at baseline, at 3 and 6 months
  The scale is measuring spasticity as response to passive movement at both slow and fast speed; scored 0 - 4. (0=no resistance; 4= inexhaustible clonus)

SECONDARY OUTCOMES:
Change in function: 5-Chair-Rise | Assessments took place at baseline, at 3 and 6 months
  The main task in this test is to get up and sit down 5 times as fast as possible without use of the arms. The goal is the global assessment of the strength of the lower limb.
Change in function: 25foot-walk-test | Assessments took place at baseline, at 3 and 6 months
  The task is to walk a 25foot distance as fast as possible. This test measures the functionality of the lower extremity and the walking speed.
Change in function: 2min-walk | Assessments took place at baseline, at 3 and 6 months
  The subject is asked to walk with the fastest, possible speed to cover the greatest possible distance in 2min.

IPD SHARING:
Plan to Share IPD: Undecided